CLINICAL TRIAL: NCT01620125
Title: Metabolic Control of Type 2 Diabetes Patients Before and After Dietary Supplementation With the Probiotic Lactobacillus Reuteri DSM 17938 - a Pilot Study
Brief Title: Metabolic Control Before and After Supplementation With Lactobacillus Reuteri DSM 17938 in Type 2 Diabetes Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Lactobacillus reuteri pilot
Record Dates: First submitted 2012-06-12; First posted 2012-06-15 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Type 2 Diabetes; Insulin Resistance
Keywords: Lactobacillus; Gut microbiota; Diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lactobacillus reuteri (Other): Dietary supplementation with Lactobacillus reuteri DSM 17938
  Interventions: Dietary Supplement: Lactobacillus reuteri DSM 17938

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri DSM 17938 — Ordinary treatment against type 2 diabetes is supplemented with one tablet containing 100 million Lactobacillus reuteri DSM 17398, once daily for 12 weeks

SUMMARY:
Recent data suggest that the trillions of bacteria in the investigators gastrointestinal tracts (gut microbiota) can function as an environmental factor that modulates the amount of body fat. Obese individuals have an altered gut microbiota and germ-free mice are resistant to developing diet-induced obesity and have lower fasting insulin and glucose and improved glucose tolerance. Administration of the probiotic bacterium Lactobacillus strain in fermented milk for 12 weeks reduced adiposity and body weight in obese adults, possibly by reducing lipid absorption and inflammatory status. However, there are no studies to the investigators knowledge that address whether probiotic supplementation improves glucose metabolism in type 2 diabetes patients.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes with a duration > 6 months
* Abdominal obesity
* HbA1c 50-80 mmol/mol
* Written informed consent
* Stated availability throughout the study period

Exclusion Criteria:

* Autoimmune diabetes eg type 1 diabetes
* Psychiatric illness or cancer diagnosis
* No foreseeable need of treatment with corticosteroids or antibiotics
* Inflammatory bowel disease
* Administration of antibiotics 4 weeks before inclusion
* Administration of probiotics 2 weeks before inclusion
* Participation in other clinical trials

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
HOMA index | 12 weeks
  To determine improved glucose handling and insulin sensitivity in adult type 2 diabetic patients supplemented with the probiotic L. reuteri DSM 17938 over a 12 week period, we assess insulin sensitivity via the HOMA index (fp-Glucose x fS-Insulin divided by 22.5).

SECONDARY OUTCOMES:
Changes in diabetes medication and hypoglycemia events | 12 weeks
  We monitor changes in diabetes medication and hypoglycemia events. Dosages of medication with oral hypoglycemic agents and number of insulin units per 24 hrs and number of hypoglycemia events will be registered in diaries.

CONTACTS AND LOCATIONS:
Overall Officials: Per-Anders E jansson, Adj prof, Principal Investigator — The Wallenberg Laboratory, Bruna Stråket 16, Sahlgrenska University Hospital S-413 45 Gothenburg, Sweden; Fredrik Bäckhed, Assoc prof, Study Chair — The Wallenberg Laboratory, Bruna Stråket 16, Sahlgrenska University Hospital, S-413 45 Gothenburg, Sweden
Locations (1):
- Gothia Forum, CTC, Gröna Stråket 12, Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Background] Backhed F, Manchester JK, Semenkovich CF, Gordon JI. Mechanisms underlying the resistance to diet-induced obesity in germ-free mice. Proc Natl Acad Sci U S A. 2007 Jan 16;104(3):979-84. doi: 10.1073/pnas.0605374104. Epub 2007 Jan 8. PMID 17210919